CLINICAL TRIAL: NCT01269242
Title: A Pilot Study to Evaluate the Efficacy and Safety of Different Bindarit Dosages in Preventing Stent Restenosis
Brief Title: The Effects of Bindarit in Preventing Stent Restenosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aziende Chimiche Riunite Angelini Francesco S.p.A (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 004SC08166; 2008-004921-40 (EudraCT Number)
Record Dates: First submitted 2011-01-03; First posted 2011-01-04 (Estimated); Last update posted 2016-08-05 (Estimated); Status verified 2016-08

CONDITIONS: Coronary Restenosis
Keywords: coronary restenosis; angioplasty; stent; MCP-1/CCL2; MCP-3/CCL7
MeSH Terms: conditions — Coronary Restenosis | interventions — bindarit

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- bindarit 600 mg (Experimental)
  Interventions: Drug: bindarit
- bindarit 1200 mg (Experimental)
  Interventions: Drug: bindarit
- placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: bindarit — 300 mg bid, that is one 300 mg tablet twice a day for 6 months;
  Arms: bindarit 600 mg
Drug: bindarit — 600 mg bid, that is two 300 mg tablets twice a day for 6 months
  Arms: bindarit 1200 mg
Drug: placebo — bindarit-matching placebo tablets for 6 months.
  Arms: placebo

SUMMARY:
The main study objective is to assess the efficacy and safety of different bindarit dosages compared to placebo in preventing restenosis, in patients submitted to coronary stenting and using a bare metal stent (Vision BMS, by Abbott).

DETAILED DESCRIPTION:
Coronary artery disease is caused by the gradual build-up of fatty deposits in coronary arteries (atherosclerosis). A diminished blood flow may cause chest pain (angina), shortness of breath or other symptoms. A complete blockage can cause a heart attack. Angioplasty and stenting techniques are safe and effective procedures performed to unblock coronary arteries. However, a recurrent problem after angioplasty is the occurrence of a new blockage, usually within 6 to 9 months after the initial procedure. This phenomenon, called "restenosis", is a body's response to the injury of the angioplasty and does not mean a progression of coronary artery disease.The pathophysiology of restenosis is complex and has as yet not been fully clarified.

Serial studies have shown that in-stent restenosis is almost exclusively caused by neointimal hyperplasia and tissue proliferation occurring in site or adjacent to the stent sites. Histological studies confirmed that neointimal hyperplasia post-stent implantation is related to vessel injury during the procedure. Chemokines have been implicated in the pathogenesis of vascular injury. In this context, MCP-1 which shows a potent chemotactic action on monocytes, can amplify the inflammatory response through the recruitment of additional monocytes. In addition, MCP-3 is known to share some key biological features with MCP-1. It has been proved that MCP-1 directly induces human vascular smooth muscle proliferation acting at this level as a potent mitogen, and that anti-MCP-1 gene therapy inhibits restenotic changes (neointimal hyperplasia) in animals after balloon injury.

An evidence of a critical increase in circulating MCP-1 after coronary angioplasty was reported. It was more evident and prolonged in patients with restenosis rather than in non-restenotic patients, in which only a transient increases in plasma MCP-1 has been demonstrated.

Since these chemokines showed to play a main role in the appearance and worsening of the restenosis process, a selective inhibitor of MCP-1 and other members of monocyte chemotactic protein subfamily of CC inflammatory chemokines (MCP-3/CCL7, MCP-2/CCL8), such as bindarit, may have a potential therapeutic use in preventing restenosis by inhibiting the VSMC proliferation, and without affecting the important process of re-endothelization.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients with no limitation of race, > 18 years of age (or minimum age as required by local regulations). Female patients of childbearing potential, required to have a negative pregnancy test and use a birth control method. Oral contraceptive are not allowed.
* Diagnosis of angina pectoris as defined by Canadian Cardiovascular Society Classification (CCS I,II, III, IV) OR unstable angina pectoris (Braunwald Classification B&C, I-II-III), or patients with documented silent ischemia.
* Maximum of two de novo lesions (>70% stenosis) per patients, to be treated with no other planned procedure within six months from the index intervention.
* Each lesion should require a single stent not longer than 28 mm and with a diameter of 2.5 mm or larger. In case additional stents are needed, the operator will be allowed to implant them in order to treat a suboptimal result such as residual edge stenosis or dissection. Additional stents should be implanted with minimal overlap. Multiple stenting should not be allowed as intention to treat strategy due to the specific inclusion criteria which has been set.
* Patients eligible for the placement of the Vision (Abbott) bare metal stent.
* The patient willing and able to cooperate with the protocol procedures, particularly attending the scheduled visits.
* Patients legally able to give written informed consent to the trial.
* A written informed consent to the trial signed and dated by the patient is available.

Exclusion Criteria:

* Patients with hypersensitivity or allergies to aspirin, heparin, clopidogrel, ticlopidine, drugs such the study medication, or any other analogue or derivative, cobalt, chromium, nickel, molybdenum or contrast media, or with a positive history for drug allergy.
* Lesions in venous or arterial grafts.
* Total occlusions.
* In-stent restenosis.
* Unprotected Left Main lesions.
* Acute myocardial infarction (ST elevation and/or Non ST Elevation) in the 48 hours prior to the procedure.
* Women with known pregnancy or who are lactating.
* Patients in whom anti-platelet and/or anticoagulation therapy is contraindicated.
* Current medical condition with a life expectancy of less than 24 months.
* The subject is participating in another device or drug study. Subject must have completed the follow-up phase of any previous study at least 30 days prior to enrolment in this trial.
* Patients under the influence of alcohol or narcotics.
* Patients with medical conditions that preclude the follow-up as defined in the protocol or that otherwise limits participation in this registry.

  m. Potassium value above the upper limit normal range.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2009-01; Primary Completion 2011-01 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
in-segment late loss (in-stent and 5 mm proximally and distally to the stent) measured by QCA | 6 months from the index procedure
  Late loss is defined as the difference between post-procedural minimum lumen diameter and 6-month minimum lumen diameter measured in-stent and in-segment.

SECONDARY OUTCOMES:
Major Adverse Cardiac Events (MACE) | 9 months
  MACE are defined as the occurrence of death, Myocardial Infarction (MI), target vessel revascularization and target lesion revascularization(CABG or PTCA).
the assessment of the safety profile of the two bindarit dosages compared to placebo | 9 months
  Safety will be assessed by monitoring the frequency of adverse events in each treatment group. Changes from baseline in physical examination, vital signs, and ECG will be also assessed. Laboratory analyses will be evaluated on the basis of the normal range, the Investigator's judgement, and mean changes from baseline (when applicable).
the imaging parameters evaluated with OCT as an optional procedure performed on a subgroup of patients. | 6 months from the index procedure
  The following parameters will be evaluated:
  * the neointimal proliferation on the surface of the stent struts;
  * the frequency of stent malapposition.
the assessment of inflammatory biomarkers in order to investigate the bindarit mechanism of action. | 9 months
  determination of the plasma levels of several circulating inflammatory biomarkers (i.e. MCP-1/CCL-2, MCP-3/CCL7) involved in the neointimal hyperplasia and tissue proliferation occurring in site or adjacent to the stent sites.

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Colombo, MD, Study Chair — Fondazione S.Raffaele del Monte Tabor - U.O Emodinamica e Cardiologia Interventistica
Locations (1):
- Fondazione S.Raffaele del Monte Tabor - UO Emodinamica e Cardiologia Interventistica, Milan, Milan, Italy

REFERENCES:
- See also: Sponsor website — http://www.angelinipharma.com